CLINICAL TRIAL: NCT04031313
Title: Effectiveness and Safety of Oil Extracts Medical Cannabis Treatment for Patients With Chronic Pain: a Web Technology Based Prospective Study
Brief Title: Effectiveness and Safety of Oil Extracts Medical Cannabis Treatment for Patients With Chronic Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dorit Pud (Other)
Collaborators: Rambam Health Care Campus (Other); Sheba Medical Center (Other Government)
Responsible Party: Sponsor-Investigator, Dorit Pud, Full Professor, University of Haifa
Organization: University of Haifa (Other)
Other Study IDs: UnivHaifa
Record Dates: First submitted 2019-07-20; First posted 2019-07-24 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: The current study will prospectively follow-up on chronic pain patients treated with oil extracts of medical cannabis (MC) for a period of six months in "real life" conditions. This study will enable a deep investigation regarding the effects of the active extract of cannabis inflorescence formulated in oil, derived from the cannabis plant. The results may allow us to reduce the gap in understanding MC's effects on pain relief and its safety, to identify predictors for treatment success/ failure, as well as to enable us tailoring a personalize MC treatment by choosing optimal concentration and dose according to the patient needs. We hypothesize that following the treatment with oil extracts of MC for chronic pain, associations will be found between its effectiveness and the types of clinical pain, personality traits and demographic characteristics. We also do not expect serious (life threatening) adverse events to be reported. Methods: This study has been already approved by the ethics committee of Haifa University (approval number 216/19). The sample will include a prospective cohort of 600 patients with chronic non-cancer pain that will request license to use oil extracts MC. The patients who will be approved to receive a license will be followed-up longitudinally for a period of six months from the signing of the consent form. The patients will be asked to fill a variety of questionnaires that may indicate the outcome of the treatment. The follow-up will take place in four time points: at the time of approval of the license (before starting the treatment, baseline), as well as at one, three, and six months from the initiation of treatment. Data will be collected by a web based data collection technology (Qualtrics®). In cases which there are a need for it, the information will be gathered by phone or face to face meetings.

DETAILED DESCRIPTION:
The use of medical cannabis (MC) for the treatment of chronic pain has risen in the last decade. According to the Israel Medical Cannabis Unit (IMCU) of the Israeli Ministry of Health (IMOH), there are currently several tens of thousands licenses for the use of medical cannabis in Israel, mostly for the relief of chronic pain (mainly utilized by smoking and inhalation). It is estimated that 2,000 new licenses will be issued yearly. Recently, the IMOH approved the use of drops of whole extract of cannabis inflorescence formulated in oil, intended for sublingual administration, for the treatment of chronic pain. That far, there is a distinct lack of evidence about the efficacy and safety of MC treatment in the long-term with relatively few prospective randomized controlled trials (RCTs) examining this issue. This can be explained, at least partially, by the reluctance of physicians, researchers and pharmaceutical companies to engage in MC research for various reasons (mainly when utilized by smoking and inhalation). Such reasons include the following facts: MC is classified as a schedule I drug by the American Food and Drug Administration (FDA); MC is often smoked; that the level of cannabinoids and terpenes can vary between suppliers and even from the same supplier and therefore it is difficult to quantify the dose; there is abuse of MC; patentability of a natural compounds is problematic; and MC consumption is stigmatized. One of the accepted ways to narrow gaps of information in medical research where there is a dearth of RCTs is to develop cohorts that may allow for the prospective, structured data collection and data mining of a large number of "real life" patient conditions.

The current study will prospectively follow-up on chronic pain patients treated with oil extracts MC for a period of six months in "real life" conditions. This study will enable a deep investigation regarding the effects of the active extract of cannabis inflorescence formulated in oil, derived from the cannabis plant. The results may allow us to reduce the gap in understanding MC's effects on pain reduction and its safety, to identify predictors for treatment success/ failure, as well as to enable us tailoring a personalize MC treatment by choosing optimal concentration and dose according to the patient needs.

Methods: The sample will include a prospective cohort of patients with chronic non-cancer pain that will request license to use oil extracts medical cannabis. The estimated sample size is 600 patients. The patients who will be approved to receive a license will be followed-up longitudinally for a period of six months from the signing of the consent form. The patients will be recruited by their physicians in their clinics.

Inclusion criteria - Patients that will be recommended to use oil extracts medical cannabis for the treatment of all forms of chronic pain (despite cancer); Patients above the age of 18 years; Patients who will sign an informed consent after receiving explanation on the requirements, duration and nature of the study.

Exclusion criteria - Patients who lack the ability to understand the purpose and instructions of the study.

Questionnaires - (1) Demographic questionnaire includes data regarding age, gender, marital status, country of origin, religion, weight, height, smoking habitats, and pain etiology; (2) Co-morbidities; (3) Expectations from cannabis treatment; (4) Information regarding the oil extracts as: type of the oil, concentration, dose, effect, etc. (5) Patient satisfaction from the treatment and the information they will be receive; (6) Pain - The short-form McGill Pain Questionnaire (SF-MPQ), Pain Disability Index (PDI), Pain treatment and other pharmacological treatments; (7) Pittsburgh Sleep Quality Index (PSQI); (8) Beck Depression Inventory (BDI-II); (9) Pain Catastrophizing Scale (PCS); (10) General Anxiety Disorder (GAD-7); (11) Quality of life (EQ5); (12) Changes in appetite; (13) Adverse events - occurrence, severity; (14) Cognitive status - by a telephone interview.

Study procedure - The study has been approved by the ethics committee of Haifa University (approval number 216/19). Participants will be recruited by physicians either with pain management expertise or those who have license to offer MC. Potential patients who will meet the inclusion criteria, will get a full explanation about the study aims and procedure. Following their agreement to participate in the study they will sign a written informed consent that will be sent to the investigator along with the patient's diagnosis and contact information. Then, the patients will be contacted by the investigator and will be asked to complete the questionnaires at each of the following time-points: at the time of approval of the license (before starting the treatment, baseline) a month, three months and six months, from the initiation of treatment. Data will be collected by a secured web based data collection technology (Qualtrics®). In case of difficulties in using that technology, the data will be collected via phone or face to face meetings. Notably, this study is only observational and not interventional, e.g., the patient will be informed that participation in this study will not influence the approval\disapproval for the acceptance\renewal of the oil extract medical cannabis license from the Medical Cannabis Unit (MCU) of the Israeli health ministry. Additionally, the research related tie between patients to their physician will be terminated following the signing of the consent form, from this point forward, the physician will have no access to the specific patients' study related data. This is in purpose to assure that decisions regarding the patient's further treatments will not be influenced by any way from the collected data.

ELIGIBILITY:
Inclusion Criteria:

* Patients that will be recommended to use oil extracts medical cannabis for the treatment of all forms of chronic pain (despite cancer)
* Patients above the age of 18 years
* Patients who will sign an informed consent after receiving explanation on the requirements, duration and nature of the study
* Only patients who will receive at least one dose of cannabis within the context of the study, will be included in the analysis.

Exclusion Criteria:

* Patients who lack the ability to understand the purpose and instructions of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample will include a prospective cohort of patients with chronic non-cancer pain that will request license to use oil extracts medical cannabis. The estimated sample size is 600 patients. The patients who will be approved to receive a license will be followed-up longitudinally for a period of six months from the signing of the consent form. The patients will be recruited by their physicians in their clinics.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in the number that best describes pain intensity during the last week (0-10) | six months
  The change from baseline in the number that best describes pain intensity during the last week (0-10)

SECONDARY OUTCOMES:
The change from baseline in PDI | six months
  The change from baseline in disability. PDI = Pain Disability Index. Total score 0-10
The change from baseline in QOL | six months
  The change from baseline in quality of life. EuroQol (EQ5). Total score 0-10
The change from baseline in SF-MPQ | six months
  The change from baseline in total McGill pain intensity score (SF-MPQ). Total score 0-45
The change from baseline in PSQI | six months
  The change from baseline in Sleep quality. Pittsburgh Sleep Quality Index (PSQI). Total score 0-21.
The change from baseline in PCS | six months
  The change from baseline in pain catastrophizing. Pain Catastrophizing Scale (PCS). Total score 0-52

CONTACTS AND LOCATIONS:
Overall Officials: Dorit Pud, PhD, Principal Investigator — University of Haifa
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No